CLINICAL TRIAL: NCT04151420
Title: Validation and Implementation of a Digital Patient Reported Remote Monitoring Tool to Systematically Monitor Mild, Moderate and Severe Infectious Complications in IBD Patients in Routine Care
Brief Title: Real Life Remote Monitoring of Mild, Moderate and Severe Infectious Complications in IBD by Patient Reported Assessment
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: MEC 2019-1115
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; IBD; Digestive System Disease; Patient Reported Outcome Measures
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult IBD patients
  Interventions: Other: Remote monitoring tool (infections questionnaire) validation

INTERVENTIONS:
Other: Remote monitoring tool (infections questionnaire) validation — There will be no treatment intervention in the current study (no drugs will be used). Instead, patients are enrolled in a routine care eHealth care-pathway with myIBDcoach. MyIBDcoach (MijnIBDcoach, Dutch, Sananet Care B.V., Sittard, The Netherlands, https://www.mijnibdcoach.nl) is a web-based platform for home-monitoring and patient- provider communication in patients with IBD.
  Patients already using the myIBDcoach will be informed on this study. Patients will be asked to continue routine care including monitoring of PROs through the myIBDcoach. When a patient completes the infections disease questionnaire for the first time, this will be regarded as the starting point (T=0) for this patient. Patients will complete the questionnaire every three months after the starting point as part of their routine follow-up. Results from these questionnaires will be stored electronically and will be analyzed alongside medical records of GP's and drug delivery data from pharmacies.

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic relapsing immune mediated inflammatory disease (IMID) of the gastrointestinal tract. Like all IMIDs (e.g. rheumatoid arthritis, psoriasis) a complex interaction between a genetically altered immune response, the gut microbiota and environmental factors is causing the disease. Systemic suppression of the immune response with corticosteroids, immunomodulatory, biologicals and combination therapies increases the risk of opportunistic infections in IBD patients.

Data on mild and moderate infections in medically treated IBD patients is scarce, mainly since infections treated by the general practitioner or in an outpatient setting are not systematically registered in real life. To help gastroenterologists with clinical decision making, real world data with long term follow-up concerning the risk for infectious complications, is warranted.

Several observations underline the importance of real world data on mild and moderate infections in medically treated IBD patients. Mild and moderate infections mostly have a benign course, but they take longer to clear and have a large impact on (work)disability and quality of life in IBD patients. Recurrent infections influences peoples willingness to use a drug and negatively effects adherence. Furthermore, recurring mild and moderate infections might prognosticate serious infections, and systematic assessment of all infections could be used to timely adjust treatment regimens and prevent serious infections.

The investigators of this study previously developed a questionnaire on self-reported infections according to the FDA guideline for patient-reported outcome measures (PROM) by interviewing 36 patients with IBD and through input of expert meetings with gastroenterologists, IBD specialists, rheumatologists, immunologists and IBD-nurses. This questionnaire has already been implemented in myIBDcoach, a validated telemedicine system implemented in routine care for over 4000 patients with IBD in the Netherlands. Assesment of reliability and validity are the last steps in validation of this remote monitoring tool.

In the current study the investigators aim to:

1. Assess the reliability, construct validity and criterion validity of a remote monitoring tool (questionnaire) for infections as last step in the validation
2. Assess the relative risk of all infections (mild, moderate and severe) in a real-life population for IBD patients on different maintenance treatments
3. Identify the predictors and risk factors of mild and moderate infections.
4. Assess the relation between patient reported infections and the risk for serious infectious complications

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and diagnosed with IBD
* Included in eHealth clinical care-pathway using myIBDcoach

Exclusion Criteria:

* Patients with insufficient knowledge of the Dutch language
* Patients not able to provide written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with medically treated inflammatory bowel disease (IBD) (ulcerative colitis and Crohn's disease) included in the eHealth clinical care-pathway using myIBDcoach and followed on the outpatient clinic of Maastricht University Medical Centre or Zuyderland Medical Centre.
Sampling Method: Non-Probability Sample
Enrollment: 584 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Remote monitoring tool validation | 24 months
  Assess the reliability, construct validity and criterion validity of a PRO for infections in IBD patients as last step in the validation.

SECONDARY OUTCOMES:
Relative risk of all infections | 12 months
  Assess the relative risk of all infections (mild, moderate and severe) in a real life population for IBD patients on different maintenance treatments
Relation between mild/moderate and serious infectious complications | 6-12 months
  Assess the relation between patient reported infections and the risk for serious infectious complications

CONTACTS AND LOCATIONS:
Overall Officials: M J Pierik, MD, PhD, Principal Investigator — Maastricht University
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Centrer, Maastricht
  - Zuyderland Medical Centre, Sittard

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to other researchers on demand. Patients will be asked to give informed consent to share the collected data with third parties for future research.
Supporting Information: Study Protocol, SAP, ICF